CLINICAL TRIAL: NCT04841772
Title: Exploring Muscle Breakdown During Exercise Recovery
Acronym: EMBER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Beachbody (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 210203-B-01
Record Dates: First submitted 2021-04-09; First posted 2021-04-12 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Muscle Damage; Healthy
Keywords: Skeletal muscle; Postabsorptive; Muscle protein breakdown; Muscle protein synthesis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegan Protein (Active Comparator)
  Interventions: Dietary Supplement: Recover Vegan Protein Supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Recover Vegan Protein Supplement — Post exercise protein supplement (26g pea protein)
  Arms: Vegan Protein
Dietary Supplement: Placebo — Post exercise placebo supplement (32g maltodextrin)
  Arms: Placebo

SUMMARY:
This study will allow researchers to explore how muscle responds to heavy exercise. The researchers will characterise rates of muscle protein breakdown and synthesis 24hours after heavy exercise with a post exercise protein polyphenol or placebo supplementation. This will inform strategies to help people recover from heavy exercise.

DETAILED DESCRIPTION:
It is well known that resistance exercise increases rates of muscle protein synthesis and breakdown, with the rise in synthesis greater in magnitude and duration. The time course of rates of muscle protein synthesis increase dramatically 24-72h following eccentric exercise, even in a non-exercised control leg. This data is consistent with a much larger increase in muscle protein breakdown than previously thought. However, the response of muscle protein breakdown following damaging eccentric exercise, and its relationship with muscle protein synthesis, has not yet been elucidated. Moreover, it is unclear whether a protein and polyphenol nutritional intervention influence rates of muscle protein breakdown to accelerate recovery. This study will allow researchers to test the hypothesis that eccentric exercise increases rates of muscle protein breakdown independently of muscle contraction per se. If this hypothesis is supported, it will highlight that recovery strategies from muscle damage should also target supporting muscle protein breakdown.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active
* 18-40 years of age

Exclusion Criteria:

* Regular and structured involvement in resistance training
* Inactive participants
* Habitual dietary protein intake <0.8g/kg bw/day and >2.0g/kg bw/day
* Regular use of nutritional supplements known to suppress inflammation or modulate protein metabolism Any diagnosed metabolic conditions (diabetes), cardiovascular disease or hypertension
* Current musculoskeletal injury
* Chronic use of anti-inflammatory medicines
* Any known disorders in muscle metabolism
* Individuals with an allergy to egg, fish, wheat or soy ingredients as the product is manufactured in a facility that contains these ingredients
* Allergy to lidocaine
* Having received or ingested a stable isotope tracer containing 15N in the past
* A personal or family history of epilepsy, seizures or schizophrenia
* Stomach bleeding or stomach ulcer
* Kidney failure
* Liver problems, such as fibrosis, cirrhosis or failure
* Crohns disease or ulcerative colitis
* Chickenpox or shingles
* Pregnant or trying to get pregnant
* Any diagnosed cardiovascular disease (e.g. deep vein thrombosis) or hypertension.
* Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes)
* Recent (within the last 6 months) or current musculoskeletal injury (leg fracture)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Muscle protein breakdown rate | 1hour
  Muscle protein breakdown rate (FBR, measured in %/h) 24hours post eccentric exercise.

SECONDARY OUTCOMES:
Muscle protein synthesis rate | 3hours
  Muscle protein synthesis rate (FSR, measured in %/h) 24hours post eccentric exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No